CLINICAL TRIAL: NCT02556333
Title: Safety and Efficacy of Emtricitabine/Tenofovir Alafenamide as Part of Salvage Antiretroviral Regimens in Patients With Uncontrolled Viremia and Drug-Resistant HIV Infection
Brief Title: Emtricitabine/Tenofovir Alafenamide as Salvage ART
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 150201; 15-I-0201 (Other: NIH)
Record Dates: First submitted 2015-09-18; First posted 2015-09-22 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-10-16

CONDITIONS: HIV
Keywords: TAF; F/TAF; antiretroviral therapy; TDF; directly observed therapy
MeSH Terms: conditions — Directly Observed Therapy | interventions — Emtricitabine; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- FTC/TAF (Experimental): Emtricitabine 200mg/tenofovir alafenamide 25mg (FTC/TAF) tablet to be given orally once daily to be added to a failing regimen for 10 days. If HIV RNA decline by >= 0.5 log copies/mL, patient will continue on FTC/TAF with a new antiretroviral regimen for 48 weeks. If < 0.5 log copies/mL decline, patient will be taken off FTC/TAF.
  Interventions: Drug: FTC/TAF

INTERVENTIONS:
Drug: FTC/TAF — Tenofovir alafenamide (TAF) is an investigational oral prodrug of tenofovir. This trial will explore the safety and efficacy of TAF in a fixed combination with emtricitabine (FTC) (F/TAF, Gilead Sciences Inc.) as part of a salvage antiretroviral regimen for HIV-1-infected adults and adolescents (greater than or equal to 14 years) who experienced virologic failure.
  Other Names: Emtricitabine 200mg/tenofovir alafenamide 25 mg (F/TAF)

SUMMARY:
Background:

HIV attacks the immune system. Antiretroviral therapy (ART) is a combination of drugs used for treating HIV infection. For some people, ART drugs stop working against their HIV. Researchers want to see if a different form of the drug tenofovir (an ART drug currently approved by the FDA), combined with another drug, may help people whose HIV is resistant to ART. This combination pill is called F/TAF

Objective:

To study the safety and efficacy of the drug F/TAF, when used with other ART, for people whose HIV infection has been hard to control with available medicines.

Eligibility:

People age 14 years and older who have HIV infection and are enrolled in the DOTCOM (14-I-0009) protocol.

Design:

Participants will be screened with physical exam, medical history, and blood and urine tests.

Participants will stay in the hospital for at least 10 days. For the first 9 days, they will take F/TAF by mouth along with their usual ART drugs.

In the hospital, they will repeat the screening tests.

Participants will have a DEXA scan, an x-ray that measures calcium and other minerals in the bones. Participants will lie on a soft table while the scanner passes over the lower spine and hips.

Participants will get a supply of F/TAF and some new ART drugs to take at home.

Participants will have follow-up visits in 1, 2, 4, 8, and 12 weeks. After the 12-week visit, they will come back about every 3 months for about 1 year.

At these visits, participants will repeat the screening tests. They will discuss any problems taking their ART drugs. They may have another DEXA scan.

DETAILED DESCRIPTION:
Despite the success of antiretroviral therapy (ART), a subset of HIV-1-infected patients have uncontrolled viremia, multiple drug class resistance, and limited treatment options. Tenofovir disoproxil fumarate (TDF) forms part of most ART regimens, however its long-term use is associated with renal tubulopathy and reduced bone mineral density. Viral mutations (eg, K65R, multiple thymidine analog mutations (TAMs) can confer resistance or reduced susceptibility to TDF.

Tenofovir alafenamide (TAF) is an investigational oral prodrug of tenofovir. When compared to TDF, TAF demonstrated lower plasma tenofovir concentrations and more potent antiviral activity at approximately one-tenth of the dose. TAF has the advantage of reduced tenofovir exposure to the renal tubules and bone, potentially resulting in fewer kidney and bone effects. As with TDF, TAF has potent activities against hepatitis B virus (HBV), and may be a treatment option for patients with HIV/HBV co-infections. Phase 2 trials have demonstrated the non-inferiority of TAF to TDF in treating HIV-1 infection in ART-naive patients. Smaller reductions in bone mineral density were measured with TAF than TDF. The most common adverse events were nausea and diarrhea.

This single-arm, single-site, open-label trial will explore the safety and efficacy of TAF in a fixed combination with emtricitabine (FTC) (F/TAF, Gilead Sciences Inc.) as part of a salvage antiretroviral regimen for HIV-1-infected adults and adolescents (greater than or equal to 14 years) who experienced virologic failure. The study will recruit patients who have failed TDF-containing regimens or cannot take TDF (due to resistance mutations or risk of renal injury) and for whom abacavir/lamivudine (ABC/3TC) is not an optimal alternative. Eligible patients will begin 9 days of inpatient directly observed therapy (DOT) with F/TAF plus their pre-enrollment background regimen. On Day 10, patients will switch to F/TAF plus OBT while waiting for the results of Day 10 HIV RNA results. Patients with an HIV RNA decline of <0.5 log10 from Day 1 to Day 10 will discontinue F/TAF, end their study participation, and continue OBT (with TDF/FTC or ABC/3TC in place of F/TAF, as appropriate) under the 14-I-0009 protocol. Patients with a greater than or equal to 0.5 log10 decline in HIV RNA will continue on F/TAF + OBT for 48 weeks, with periodic outpatient assessments of adherence, safety, renal function, bone mineral density, HIV RNA, and CD4 T cell counts. Switching of one or more drugs in an ART regimen due to inadequate viral response will require inpatient DOT under 14-I-0009.

ELIGIBILITY:
INCLUSION

* Age greater than or equal to 14 years
* Documented HIV-1 infection (written documentation of positive standard ELISA or rapid HIV-1/HIV-2 antibody test with confirmatory Western Blot, or documentation of repeated HIV RNA of > 1,000 copies/mL)
* Concurrent enrollment in the DOTCOM (14-I-0009) protocol
* For females of childbearing potential, willingness to use effective contraception for the duration of the study
* Willingness to be hospitalized for 10-15 days (with potential for day passes)
* Willingness to have blood samples stored for future research that may include genetic testing
* Multiple ART failure as defined by at least one of the following criteria:

  * HIV RNA > 1000 copies/mL and documented virologic failure on at least 1 prior ART regimen and at least 2 consecutive HIV RNA plasma measurements of > 1,000 copies/mL, including the last documented value, while on the currently prescribed ART regimen for at least 6 months; or
  * Documented extensive resistance to at least 3 antiretroviral (ARV) drug classes, and persistent plasma viremia (HIV RNA > 1,000 copies/mL for > 6 months) despite multiple regimen changes. The patient may be enrolled even if they have been prescribed their current regimens for less than 6 months.
* Where neither TDF nor ABC are optimal NRTI options as defined by at least one of the following criteria:

  * Presence of the M184V mutation plus TDF-associated resistance mutations based on genotypic/phenotypic testing, specifically K65R alone, or with TAMs (such as 41L, 67N, 70R, 210W, 215Y/F, or 219Q/E) with or without other NRTI-associated mutations; or
  * FTC/TDF is not considered an option due to impaired renal function (eGFR by Cockroft-Gault equation [eGFR(CG)]=30-60 mL/min), or risk of renal impairment because of conditions such as uncontrolled hypertension, diabetes mellitus, or history of renal toxicity while receiving a TDF-based regimen; and where ABC/3TC is contraindicated (ie, presence of HLA B*5701 allele or history of hypersensitivity reaction to ABC), or is a suboptimal option (eg, presence of ABC-associated resistance mutation(s) or in patients with HBV co-infection).

EXCLUSION

* Severe renal impairment (eGFR(CG) <30 mL/min)
* Acute medical illness stemming from a significant co-morbidity (eg, malignancy requiring chemotherapy, treatment of an acute opportunistic infection or acute renal failture). Enrollment may be deferred up to 3 months to allow a condition to resolve or stabilize.
* Pregnancy; however if a patient becomes pregnant while enrolled in the protocol, she may continue participation throughout her pregnancy.
* Breastfeeding
* Concomitant use of one of the following medications: carbamazepine, oxcarbazepine, phenobarbital, phenytoin, rifabutin, rifampin, rifapentine, bisphosphonate, St. John s wort, echinacea, milk thistle, sho-saiko-to, and probenecid.
* Any illness or condition that, in the investigator's opinion, may substantially increase the risk of participation in the study, or compromise the scientific objectives.

Ages: 14 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-09-16; Primary Completion 2016-08-16 (Actual); Study Completion 2016-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Pau, Pharm.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dombrowski JC, Kitahata MM, Van Rompaey SE, Crane HM, Mugavero MJ, Eron JJ, Boswell SL, Rodriguez B, Mathews WC, Martin JN, Moore RD, Golden MR. High levels of antiretroviral use and viral suppression among persons in HIV care in the United States, 2010. J Acquir Immune Defic Syndr. 2013 Jul 1;63(3):299-306. doi: 10.1097/QAI.0b013e3182945bc7. PMID 23572013
- [Background] Deeks SG, Gange SJ, Kitahata MM, Saag MS, Justice AC, Hogg RS, Eron JJ, Brooks JT, Rourke SB, Gill MJ, Bosch RJ, Benson CA, Collier AC, Martin JN, Klein MB, Jacobson LP, Rodriguez B, Sterling TR, Kirk GD, Napravnik S, Rachlis AR, Calzavara LM, Horberg MA, Silverberg MJ, Gebo KA, Kushel MB, Goedert JJ, McKaig RG, Moore RD. Trends in multidrug treatment failure and subsequent mortality among antiretroviral therapy-experienced patients with HIV infection in North America. Clin Infect Dis. 2009 Nov 15;49(10):1582-90. doi: 10.1086/644768. PMID 19845473
- [Background] Ezinga M, Wetzels JF, Bosch ME, van der Ven AJ, Burger DM. Long-term treatment with tenofovir: prevalence of kidney tubular dysfunction and its association with tenofovir plasma concentration. Antivir Ther. 2014;19(8):765-71. doi: 10.3851/IMP2761. Epub 2014 Feb 28. PMID 24584104

RESULTS

PARTICIPANT FLOW:
Groups:
- TAF Treatment: Each subject receives tenofovir alafenamide (TAF) with emtricitabine to be added to a failing antiretroviral regimen for 10 days, if there is a HIV RNA response of >= 0.5 log decline, subjects will continue of TAF with emtricitabine with a new optimized background regimen. If <0.5 log decline, TAF with emtricitabine will be discontinued and study enrollment for the subject will be terminated.
Period: Overall Study
Arm/Group | TAF Treatment
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | TAF Treatment
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: HIV RNA Change From Baseline to Day 10
Description: An HIV RNA decline of >=0.5 log by day 10 will be considered to be an adequate virologic response, to proceed to the second phase of the study.
Time Frame: 10 days
Population: One patient with multiple drug resistant HIV infection enrolled into this study.
Measure: Number; unit: log HIV RNA copies/mL
Arm/Group | TAF Treatment
Number analyzed (Participants) | 1
log HIV RNA copies/mL | 0.01

ADVERSE EVENTS:
Time Frame: 10 days
Arm/Group | TAF Treatment
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
The study was approved in late 2015, with the first and only patient enrolled in Jan 2016. The drug was approved in April 2016, which resulted in termination of the protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2015-09-02): https://cdn.clinicaltrials.gov/large-docs/33/NCT02556333/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2015-08-31): https://cdn.clinicaltrials.gov/large-docs/33/NCT02556333/Prot_SAP_002.pdf